CLINICAL TRIAL: NCT02661802
Title: Acute Effects of 40% Oxygen Supplementation Determined Better Exercise Capacity in Eisenmenger Syndrome
Brief Title: Effects Oxygen Supplementation Determined Better Exercise Capacity in Eisenmenger Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Laion rodrigo do Amaral Gonzaga, Principal Investigator, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13473813.1.0000.5505
Record Dates: First submitted 2016-01-20; First posted 2016-01-22 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Eisenmenger Complex; Hypertension, Pulmonary
MeSH Terms: conditions — Eisenmenger Complex; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxygen Supplementation (Experimental): Two six-minute walk tests, one with oxygen supplementation and another without were performed on different days. During the test with oxygen supplementation the delivery was continuous by mask at 40% and technician walked behind the patient with the oxygen source.
  Interventions: Other: Oxygen Supplementation

INTERVENTIONS:
Other: Oxygen Supplementation — Oxygen delivery was continuous by mask at 40%

SUMMARY:
The purpose of this study was to evaluate the acute effects of oxygen supplementation during a submaximal exercise test in patients with Eisenmenger's Syndrome.

DETAILED DESCRIPTION:
Patients with Eisenmenger's syndrome were submitted to a submaximal exercise test (six-minute walking test) with and without supplemental oxygen. The distance walked during the two tests were compared to assess the impact of oxygen supplementation on the walking distance.

ELIGIBILITY:
Inclusion Criteria:

* Abscence of heart failure and/or respiratory infection
* Advanced therapy for pulmonary hypertension

Exclusion Criteria:

* Lung, liver or connective tissue diseases
* Neuromuscular diseases
* Inability to perform a pulmonary function test and/or chronic lung disease
* Inability to walk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Distance walked during the six-minute walk tests | At enrollment
  Distance walked during the six-minute walk tests with and without oxygen supplementation were recorded and compared to each other to establish the impact of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laion Gonzaga, PT, Principal Investigator — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared. However, all enrolled subjects were provided the principal investigator's phone number and e-mail address in order to receive test results and ask questions.